CLINICAL TRIAL: NCT02136719
Title: Bimanual Uterine Compression to Reduce Blood Loss and Prevent Postpartum Haemorrhage After Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: khalidkhader 2
Record Dates: First submitted 2014-05-11; First posted 2014-05-13 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Postpartum Haemorrhage
Keywords: Uterine massage; vaginal birth; postpartum haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): bimanual uterine compression immediately after delivery of placenta for 5 minutes in 260 women
  Interventions: Procedure: bimanual uterine compression
- Group B (No Intervention): no intervention (260 women).

INTERVENTIONS:
Procedure: bimanual uterine compression — bimanual uterine compression immediately after delivery of placenta for 5 minutes
  Arms: Group A

SUMMARY:
the investigators aim to compare bimanual uterine compression immediately after delivery of the placenta for 5 minutes versus no intervention for the prevention of postpartum hemorrhage in Women at high risk for primary atonic postpartum hemorrhage. The primary outcome is postpartum haemorrhage (blood loss of ≥ 500 ml) while the Secondary outcomes include use of additional uterotonics and need for blood transfusion.

DETAILED DESCRIPTION:
the investigators conduct a prospective non- randomized study at Department of Obstetrics and Gynecology, Benha University Hospital, since April 2014 till May 2016, after approval of the study protocol by the Local Ethical Committee. A written informed consent is obtained from eligible women before induction or at early stage of labour.

Women with singleton pregnancies of more than 28 weeks' gestation who are admitted to hospital and candidates for vaginal delivery are eligible for the study .Gestational age more than 28 weeks the gestational age is determined based upon the date of the first day of last normal menstrual period and confirmed by ultrasound scan during the 1st trimester.

The patients (520) are divided into two groups, Group A (260) receive bimanual uterine compression immediately after delivery of the placenta for 5 minutes while Group B (260) receive no intervention.

The third stage of labour was managed as usual by clamping and cutting of umbilical cord, waiting for signs of placental separation and delivering the placenta by controlled cord traction.

Duration of the 3rd stage of labour is calculated. Patients are kept in labor room under observation for a period of 1 h.

Measurement of blood loss by a clean plastic lined absorbent drape placed under the woman's buttocks to collect all the blood lost after delivery of the baby and drainage of the amniotic fluid. The drape is changed as many times as needed. The woman stays on the drape or asked to wear a pad over the next 60 minutes. In the case of severe haemorrhage, the investigators follow the usual guidelines for management of postpartum haemorrhage, and the supplemental treatment registered. All drapes and pads are weighed on an electronic scale and the known dry weight of the linen is subtracted. As 1 ml of blood weighs close to 1 g, the balance in grams is assumed to be the total blood loss in ml.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age more than 28 weeks the gestational age was determined based upon the date of the first day of last normal menstrual period and confirmed by ultrasound scan during the 1st trimester
2. Women at high risk for primary atonic postpartum hemorrhage

   * Over distended uterus
   * Large fetus
   * Multiple fetuses
   * Hydramnios
   * Distension with clots accidental hemorrhage
   * Exhausted myometrium
   * Prolonged labor
   * Oxytocin or prostaglandin stimulation
   * Chorioamnionitis
   * Previous uterine atony
   * Placenta previa
   * Marked anemia

Exclusion Criteria:

1. Cervical tear
2. extensive birth canal tear
3. Postpartum hemorrhage
4. Retained placenta
5. Coagulopathy
6. Chronic medical illness hepatic renal
7. Pregnancy induced hypertension PIH
8. Refusal to participate in the study

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss 500 ml or more after enrolment | 60 minutes after enrolment
  estimating blood loss from vagina

SECONDARY OUTCOMES:
Blood loss 1000 ml or more after enrolment | (up to 30 and 60 minutes) after enrolment
  estimating blood loss by collecting it
Use of additional uterotonics or other procedures | 60 minutes
  giving drugs IV
Blood transfusion | 60 minutes
  giving how many units of PRBCS

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim zweel, Principal Investigator — Department of Obstetrics and Gynecology,AFHSA
Locations (1):
- Benha univesity hospital and afhsa, Banhā, El Qualyobia, Egypt